CLINICAL TRIAL: NCT00869804
Title: Pilot Randomized Study of Aerobic and Resistance Exercise for Women Undergoing Treatment for Breast Cancer With Taxanes.
Brief Title: Heading Off Peripheral Neuropathy With Exercise
Acronym: HOPE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not recruit total numbers needed. PI left institution.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0478-08-FB
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Nervous System Disorders; Breast Neoplasms; Chemotherapy
Keywords: breast cancer; chemotherapy-induced peripheral neuropathy; exercise
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): combination aerobic (walking) and resistance (strength training) exercise
  Interventions: Behavioral: Aerobic/ Resistance Exercise Intervention
- attention control (Sham Comparator): attention control with daily journal and cancer-related education
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: Aerobic/ Resistance Exercise Intervention — The intervention will consist of a tailored home-based program of both aerobic (walking, using pedometer) and strength training exercises for upper and lower extremities using resistance power bands.
  Arms: Exercise
Behavioral: Attention control
  Arms: attention control

SUMMARY:
Chemotherapy for the treatment of breast cancer can affect nerves and muscles leading to loss of sensation in the hands and feet for feeling hot and cold, difficulty walking, and muscle weakness. This study will explore if exercises such as walking and strength training may prove helpful in preventing or lessening chemotherapy-induced peripheral neuropathy from chemotherapy, making the therapy easier to tolerate and increasing overall quality of life.

DETAILED DESCRIPTION:
This pilot study will test the effects of a tailored home-based walking (aerobic) and strength training (resistance) exercise program for individuals receiving taxane-based chemotherapy for breast cancer on neuropathy, breast cancer-related symptoms, cold thermal sensation, vibratory sensation, gait & balance, upper and lower extremity muscle strength, and quality of life.

The objective of this pilot study is to determine the effect size, feasibility and acceptability of a 12-week combination exercise program consisting of aerobic exercise (walking) and strength training for preventing or ameliorating the clinical manifestations and symptoms of CIPN in individuals with Stage I-IIIa non-metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* age 19 or older with newly diagnosed Stage I-IIIa invasive breast cancer who are to be treated with a taxane-based chemotherapy regimen (with paclitaxel or docetaxel) and thus are at risk for the development of CIPN.

Exclusion Criteria:

* any disease (e.g. diabetes, HIV) that results in peripheral neuropathy;
* any disease or disorder that results in muscle weakness (such as chronic fatigue syndrome, multiple sclerosis, spinal cord tumors or injuries, stroke, preexisting cardiopulmonary disease);
* any disease or disorder that would preclude strength training exercises (such as bone metastasis, osteoporosis);
* individuals with diagnosed lymphedema or advanced disease (> Stage IIIa, or metastatic disease) at high risk for bone metastases and pathologic fracture will be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-03-25 (Actual); Primary Completion 2011-12-13 (Actual); Study Completion 2011-12-13 (Actual)

PRIMARY OUTCOMES:
effect size for reduction of neuropathic symptoms | Baseline, 4, 8 12, 24 weeks
  effect size for reduction of neuropathic symptoms

SECONDARY OUTCOMES:
effect size for potential covariates on measures of chemotherapy-induced peripheral neuropathy | Baseline, 4, 8, 12, 24 weeks
  effect size for potential covariates (age, taxane dose, baseline level of exercise participation, breast cancer-related symptoms) on measures of chemotherapy-induced peripheral neuropathy
feasibility and acceptability of a home-based aerobic and strength training exercise program | Baseline, 4, 8, 12, 24 weeks
  determine the feasibility and acceptability of a home-based aerobic and strength training exercise program during and after taxane-based chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Constance Visovsky, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States